CLINICAL TRIAL: NCT00184262
Title: Exposure and Response Prevention (ERP) With Behavioral- Versus Cognitive Therapy Rationale in the Treatment of OCD
Brief Title: Exposure and Response Prevention With Behavioral- Versus Cognitive Therapy Rationale in Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4941.1
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy; Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERP cognitive therapy (Active Comparator)
  Interventions: Behavioral: ERP cognitive therapy
- ERP behavioral therapy (Experimental)
  Interventions: Behavioral: ERP behavioral therapy

INTERVENTIONS:
Behavioral: ERP cognitive therapy — 15 exposure and response prevention (ERP) sessions in 3 months with a cognitive therapy rationale
  Other Names: exposure and response prevention + cognitive therapy
  Arms: ERP cognitive therapy
Behavioral: ERP behavioral therapy — 15 exposure and response prevention (ERP) sessions in 3 months with a behavioral therapy rationale
  Other Names: exposure and response prevention + behavioral therapy
  Arms: ERP behavioral therapy

SUMMARY:
The aim of the study is to determine whether exposure and response prevention (ERP) is more effective when patients are presented with a behavioral therapy versus cognitive therapy rationale in the treatment of obsessive-compulsive disorder (OCD).

DETAILED DESCRIPTION:
The aim of the study is to determine whether exposure and response prevention (ERP) is more effective when patients are presented with a behavioral therapy versus cognitive therapy rationale in the treatment of obsessive-compulsive disorder OCD.

A randomized controlled trial including patients with OCD. 50 patients will receive 15 ERP sessions in 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Obsessive-compulsive disorder

Exclusion Criteria:

* active thought disorder, uncontrolled bipolar disorder, mental retardation, organic mental disorder, initiation or change in medication three months prior to inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2003-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
scores on Y-BOCS and SCID-I | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: K. Gunnar Götestam, PhD MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, INM, Trondheim, Norway

REFERENCES:
- [Result] Hansen B, Vogel PA, Stiles TC, Gotestam KG. Influence of co-morbid generalized anxiety disorder, panic disorder and personality disorders on the outcome of cognitive behavioural treatment of obsessive-compulsive disorder. Cogn Behav Ther. 2007;36(3):145-55. doi: 10.1080/16506070701259374. PMID 17943480